CLINICAL TRIAL: NCT05243719
Title: An Open-Label Extension Study Evaluating the Safety and Efficacy of ADP101 for Oral Immunotherapy in Food-Allergic Children and Adults (The Encore Study)
Brief Title: Open-label Extension Study of ADP101
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Alladapt Immunotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADP101-MA-02
Record Dates: First submitted 2022-02-03; First posted 2022-02-17 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Food Allergy
Keywords: ADP101; Allergy; Oral immunotherapy; OIT; Allergies; Food allergies; Multi-food allergic; Multi-allergen oral immunotherapy; Tree nut allergy; Milk allergy; Wheat allergy; Egg allergy; Fin fish allergy; Shrimp allergy; Peanut allergy; Sesame seed allergy; Soy allergy; Shellfish allergy; Fish allergy; Seafood allergy; Dairy allergy; Desensitization; Food hypersensitivity; Immune system disease; Hypersensitivity, immediate; Hypersensitivity
MeSH Terms: conditions — Food Hypersensitivity; Hypersensitivity; Nut Hypersensitivity; Milk Hypersensitivity; Wheat Hypersensitivity; Egg Hypersensitivity; Peanut Hypersensitivity; Shellfish Hypersensitivity; Immune System Diseases; Hypersensitivity, Immediate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Options 1, 2, 3, 4, 5 (Experimental): Participants will fall into 1 of 5 treatment options dependent on the treatment received (ADP101 or placebo) during the parent study and their tolerance of the treatment regimen during the parent study.
  Interventions: Biological: ADP101

INTERVENTIONS:
Biological: ADP101 — Active dry powder formulation at various volumes.

SUMMARY:
This is an open-label, safety extension study for participants who participated in the Harmony study (protocol ADP101-MA-01).

DETAILED DESCRIPTION:
This study is enrolling participants by invitation only. This is a multicenter, open-label, long-term extension study of the safety and efficacy of ADP101 for oral immunotherapy in food allergic children and adults who completed the Harmony study (protocol ADP101-MA-01).

ELIGIBILITY:
Key Inclusion Criteria:

• Subjects must have completed the ADP101-MA-01 (The Harmony Study) and been compliant with study drug per protocol

Key Exclusion Criteria:

* History of or current EoE, other eosinophilic gastrointestinal disease, chronic, recurrent or severe GERD, symptoms of dysphagia
* Hypersensitivity to epinephrine or any of the excipients in ADP101
* Prior or concurrent therapies as follows:

  * beta-blockers, ACE inhibitors, ARBs or calcium channel blockers
  * regular steroid medication use
  * therapeutic antibody treatment currently or within the previous 6 months
  * any food immunotherapy currently or within the previous 12 weeks, except ADP101
  * investigational agents other than ADP101
  * in the build up phase of non-food immunotherapy
* Any other condition that might preclude safe participation in the study

Ages: 4 Years to 57 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-02-27 (Actual)

PRIMARY OUTCOMES:
Long-term safety and tolerability of ADP101 | Through study completion, approximately 4-6 years
  Incidence of adverse events including serious adverse events during the study period.

SECONDARY OUTCOMES:
Food Allergy Desensitization | Week 40
  The proportion of subjects who tolerate a highest dose of at least 600-mg level of protein from a relevant allergen or allergens without dose-limiting symptoms at the Week 40 double-blind placebo-controlled food challenge.

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Lun Wang, MD, Study Director — VP of Clinical Development, Alladapt Immunotherapeutics, Inc.
Locations (14):
- United States (14):
  - Study Site, Mission Viejo, California
  - Study Site, Rolling Hills Estates, California
  - Study Site, San Diego, California
  - Study Site, Colorado Springs, Colorado
  - Study Site, Denver, Colorado
  - Study Site, Tampa, Florida
  - Study Site, Atlanta, Georgia
  - Study Site, Marietta, Georgia
  - Study Site, Normal, Illinois
  - Study Site, Ann Arbor, Michigan
  - Study Site, Chapel Hill, North Carolina
  - Study Site, Cincinnati, Ohio
  - Study Site, Charleston, South Carolina
  - Study Site, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No